CLINICAL TRIAL: NCT02974816
Title: The Glooko Diabetes Mobile Monitoring and Management Advantage Study
Brief Title: Glooko mHealth Advantage Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glooko (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL1
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Glooko; Mobile health application; Insulin treated; Type 2 Diabetes; Remote patient monitoring; Certified diabetes educator; mHealth Advantage; Population health
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Subjects in this arm will visit their physician once every 3 months and will receive usual care.
- Remote Monitoring (Experimental): Subjects in this arm will visit their physician once every 3 months and will receive usual care. In addition, in between clinic visits, subjects will measure their blood glucose (BG) readings at least once a day and share their BG readings with their CDE using Glooko's mobile application. Once a week, the CDE will review the subject's BG readings on Glooko's population tracker and reach out to the subjects if he/she experienced clinical incident(s). During the conversation, the CDE will either recommend medication or lifestyle modification to address the clinical incident.
  Interventions: Device: Glooko's mobile application

INTERVENTIONS:
Device: Glooko's mobile application — Standard of care and Remote monitoring
  Other Names: Glooko's Population Tracker, Meter Sync Blue
  Arms: Remote Monitoring

SUMMARY:
The purpose of this study is to compare HbA1c of insulin-treated subjects with type 2 diabetes managed via usual care alone and usual care augmented with remote monitoring using Glooko

DETAILED DESCRIPTION:
In this study, the investigator wants to evaluate if diabetes self-management supported by a mobile application, which captures a subject's blood glucose readings, lifestyle and medication information and shares it with the subject's certified diabetes educator (CDE) to enable remote monitoring, improves their glycemic control compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act (HIPAA) or other privacy authorization prior to any participation in study.
2. Subject has self-reported type 2 diabetes.
3. Subject has HbA1c ≥ 7.5% and ≤ 12.5% measured within 30 days of screening visit.
4. Subject is on a stable diabetes therapeutic regimen of two or more diabetic medications (e.g., metformin plus one other antihyperglycemic agent) and/or insulin therapy for at least 2 months before screening visit. Dose changes or adjustments made within 2 months is acceptable as long as the patient has been on the medication regimen for 2 months or longer.
5. Subject is ≥ 18 and ≤ 75 years of age.
6. Subject is a male or non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit. A urine pregnancy test is required for all female subjects unless she is not of childbearing potential, defined as postmenopausal for at least one year prior to screening visit or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
7. If female is of childbearing potential, is practicing one of the following methods of birth control (and will continue through the duration of the study):

   1. Condoms, sponge, diaphragm, or intrauterine device;
   2. Oral or parenteral contraceptives for 3 months prior to screening visit;
   3. Vasectomized partner;
   4. Total abstinence from sexual intercourse
8. Subject is able to speak, read and write in English
9. Subject has a Glooko compatible smartphone/device with an active data plan or access to Wi-Fi and downloaded at least one mobile application on their phone on their own.
10. Subject has performed self-monitoring of blood glucose at least five (5) times within two (2) weeks prior to screening visit.

Exclusion Criteria:

1. Subject has type 1 diabetes.
2. Subject has advanced disease (physical or psychological) that would prevent them from being able to comply with study tasks and considered exclusionary by the study physicians.
3. Subject has been on medication or therapy within the last 2 months that severely affects blood glucose levels (e.g. corticosteroids).
4. Subject has visual impairment which severely limits his/her ability to see or use the mobile application.
5. Subject is a participant in another clinical study that has not been approved as a concomitant study by Glooko.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | 24 weeks
  Change in HbA1c from baseline

SECONDARY OUTCOMES:
Change in HbA1c from baseline | 12 weeks
  Change in HbA1c from baseline
Percentage of patients achieving </=7% | 12 and 24 weeks
  Percentage of patients achieving </=7%
Basal insulin dose(Change from baseline) | 12 and 24 weeks
  Basal insulin dose(Change from baseline)
Bolus insulin dose(Change from baseline) | 12 and 24 weeks
  Bolus insulin dose(Change from baseline)
Change in Total insulin dose(Change from baseline) | 12 and 24 weeks
  Change in Total insulin dose(Change from baseline)
Weight(Change from baseline) | 12 and 24 weeks
  Weight(Change from baseline)
Problem Areas in Diabetes score(Change from baseline) | 12 and 24 weeks
  Problem Areas in Diabetes score(Change from baseline)
Rate of hypoglycemic events (blood glucose level <70mg/dL) | 12 and 24 weeks
  Rate of hypoglycemic events (blood glucose level <70mg/dL)
Self-monitoring blood glucose frequency | 12 and 24 weeks
  Self-monitoring blood glucose frequency
Mean blood glucose concentration(Change from baseline) | 12 and 24 weeks
  Mean blood glucose concentration(Change from baseline)
Number of ER visits(Change from baseline) | 12 and 24 weeks
  Number of ER visits(Change from baseline)
Number of hospitalizations(Change from baseline) | 12 and 24 weeks
  Number of hospitalizations(Change from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Greenfield, MD, Study Director — Glooko
Locations (4):
- United States (4):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Sutter Health, Elk Grove, California
  - Scripps Whittier Diabetes Institute, San Diego, California
  - Billings Clinic, Billings, Montana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang ES, Basu A, O'Grady M, Capretta JC. Projecting the future diabetes population size and related costs for the U.S. Diabetes Care. 2009 Dec;32(12):2225-9. doi: 10.2337/dc09-0459. PMID 19940225
- [Background] Cowie CC, Rust KF, Ford ES, Eberhardt MS, Byrd-Holt DD, Li C, Williams DE, Gregg EW, Bainbridge KE, Saydah SH, Geiss LS. Full accounting of diabetes and pre-diabetes in the U.S. population in 1988-1994 and 2005-2006. Diabetes Care. 2009 Feb;32(2):287-94. doi: 10.2337/dc08-1296. Epub 2008 Nov 18. PMID 19017771
- [Background] Quinn CC, Shardell MD, Terrin ML, Barr EA, Ballew SH, Gruber-Baldini AL. Cluster-randomized trial of a mobile phone personalized behavioral intervention for blood glucose control. Diabetes Care. 2011 Sep;34(9):1934-42. doi: 10.2337/dc11-0366. Epub 2011 Jul 25. PMID 21788632
- [Background] Standards of medical care in diabetes--2015: summary of revisions. Diabetes Care. 2015 Jan;38 Suppl:S4. doi: 10.2337/dc15-S003. No abstract available. PMID 25537706
- [Background] Fisher L, Glasgow RE, Mullan JT, Skaff MM, Polonsky WH. Development of a brief diabetes distress screening instrument. Ann Fam Med. 2008 May-Jun;6(3):246-52. doi: 10.1370/afm.842. PMID 18474888
- [Background] Welch GW, Jacobson AM, Polonsky WH. The Problem Areas in Diabetes Scale. An evaluation of its clinical utility. Diabetes Care. 1997 May;20(5):760-6. doi: 10.2337/diacare.20.5.760. PMID 9135939
- [Background] UK Prospective Diabetes Study Group. Tight blood pressure control and risk of macrovascular and microvascular complications in type 2 diabetes: UKPDS 38. UK Prospective Diabetes Study Group. BMJ. 1998 Sep 12;317(7160):703-13. PMID 9732337
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. in 2012. Diabetes Care. 2013 Apr;36(4):1033-46. doi: 10.2337/dc12-2625. Epub 2013 Mar 6. PMID 23468086